CLINICAL TRIAL: NCT00469040
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, 14 Day Repeat Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Extra-pulmonary Pharmacodynamics of Inhaled Doses of GW642444M Formulated With Magnesium Stearate in Healthy Subjects
Brief Title: Safety, Blood Levels and Effects of GW642444
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2C108784
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GW642444,; healthy subjects; magnesium stearate,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- GW642444M 25mcg (Experimental): In Cohort 1 if subjects meet the stopping criteria the dose of GW642444M will changed to one inhalation of 25 mcg.
  Interventions: Drug: GW642444M for 14 days
- GW642444M 50mcg (Experimental): Subjects after randomization will receive two inhalations of 25 mcg GW642444M in Cohort 1.
  Interventions: Drug: GW642444M for 14 days
- GW642444M 100mcg (Experimental): In Cohort 2 if subjects meet the stopping criteria the dose of GW642444M will changed to one inhalation of 100 mcg.
  Interventions: Drug: GW642444M for 14 days
- GW642444M 200mcg (Experimental): Subjects after randomization will receive two inhalations of 100 mcg GW642444M in Cohort 2.
  Interventions: Drug: GW642444M for 14 days
- GW642444M 400mcg (Experimental): Subjects after randomization will receive two inhalations of 200 mcg GW642444M in Cohort 3.
  Interventions: Drug: GW642444M for 14 days

INTERVENTIONS:
Drug: GW642444M for 14 days — M salt
  Other Names: GW642444 (25; 50; 100; 200 & 400 mcg) for 14 days

SUMMARY:
GW642444 (the study medicine) is a new experimental medicine for treating asthma and chronic obstructive pulmonary disease (COPD). People with asthma and COPD suffer from breathlessness because the small tubes (bronchioles) that carry air in and out of the lungs become narrow. We hope that the study medicine will work by relaxing the muscles in the airways and help to keep the airways open, and make breathing easier. The study medicine might improve on available treatments by having fewer side-effects, and by working faster and for longer, so that patients could take it once daily, instead of twice daily.

When a medicine is made into a form ready to be given to patients, inactive ingredients are often added. Inactive ingredients might be used to help a medicine work better, to make it easier to produce the medicine, or to make it easier to get an accurate dose of medicine. In this study, the study medicine contains the inactive ingredient magnesium stearate.

We need to check that the study medicine doesn't cause problems when inhaled along with magnesium stearate. So, we're doing this study in healthy people to find out the answers to these questions.

1)Do repeated once-daily doses of the study medicine cause any important side effects when inhaled, along with magnesium stearate, as a fine powder? 2)How much of the study medicine gets into the bloodstream and how long does the body take to get rid of it?

ELIGIBILITY:
Inclusion criteria:

* healthy males and females (of non-childbearing potential) aged 18-55
* body weight >50kg with BMI 19-29.9 kg/m2
* normal ECG recording
* non-smoker

Exclusion criteria:

* high blood pressure (above 140/90 mmHg)
* pulse outside range 45 - 90 bpm
* history of breathing problems e.g. asthma
* low haemoglobin (<11 g/dL)
* blood donation within 56 days of study start
* taking regular medication
* participation in another trial within 4 months of study start
* history of drug or alcohol abuse
* abnormal clinical laboratory tests
* known allergies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-02-28 (Actual); Primary Completion 2007-04-16 (Actual); Study Completion 2007-04-16 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability as measured by ECG, blood pressure, pulse rate and blood and urine tests. Repeated measures on Day 1, 7 and 14 | Repeated measures on Day 1, 7 and 14

SECONDARY OUTCOMES:
Effects of the medicine on the body as measured by potassium and glucose levels in the blood. Monitoring of the study medicine in the body by analysis of blood samples. Repeated measures on Day 1, 7 and 14 | Repeated measures on Day 1, 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kempsford R, Norris V, Siederer S. Vilanterol trifenatate, a novel inhaled long-acting beta2 adrenoceptor agonist, is well tolerated in healthy subjects and demonstrates prolonged bronchodilation in subjects with asthma and COPD. Pulm Pharmacol Ther. 2013 Apr;26(2):256-64. doi: 10.1016/j.pupt.2012.12.001. Epub 2012 Dec 8. PMID 23232038
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study B2C108784 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/B2C108784?search=study&search_terms=B2C108784#rs
- Available data/document: Statistical Analysis Plan: B2C108784 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C108784 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2C108784 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C108784 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2C108784 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C108784 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C108784 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register